CLINICAL TRIAL: NCT00846313
Title: A Randomised Study of Dietary Counseling for Patients With Colorectal Cancer.
Brief Title: Can Malnutrition be Prevented in Patient With Colorectal Cancer Stage Dukes D?
Acronym: ColErn
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was stopped due to lack of resources (clinical dietitians)
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2002.127; 10641 (Other: The Data Inspectorate); 03/05111 (Other: Biobank)
Record Dates: First submitted 2009-02-16; First posted 2009-02-18 (Estimated); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Colorectal Neoplasm
Keywords: Dietary intake; Dietary counseling; Weight loss; Body composition; Resting energy expenditure; Quality of life
MeSH Terms: conditions — Colorectal Neoplasms; Weight Loss | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dietary counseling (Active Comparator): Patients receive dietary advice at an individual level and are offered contact with clinical dietitian every second week if necessary.
  Interventions: Other: Individual dietary counseling.
- Control (No Intervention)

INTERVENTIONS:
Other: Individual dietary counseling. — Dietary advice based on individual requirement and symptom burden. Dietary intervention may be dietary advice, energy rich foods and drinks, oral nutritional supplements, appetite stimulation with Megestrol Acetate, enteral or parenteral nutrition.
  Other Names: Dietary intervention.
  Arms: Dietary counseling

SUMMARY:
The purpose of this randomised intervention study is to investigate to what degree patients with colorectal cancer benefit of dietary counselling regarding nutritional status, oncologic treatment and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* metastatic colorectal cancer
* histological verified cancer
* age >18 years

Exclusion Criteria:

* cognitive reduction
* confusion
* not able to answer questionaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2003-12; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Body weight | 2 year

SECONDARY OUTCOMES:
Body composition | 2 year
Quality of life | 2 years
Oncologic treatment | 2 years
Dietary intake | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Lene Thoresen, MSc, Principal Investigator — St. Olavs Hospital, NTNU